CLINICAL TRIAL: NCT04192513
Title: A Randomized, Observer-Blinded, Vehicle Controlled, Single Dose, Dose Escalating, Single Application Within-patient Bilateral Comparison to Study the Safety and Antimicrobial Efficacy of DBI-001 Gel Vs. Placebo
Brief Title: Observer-Blinded Dose Escalating, Single Dose to Study Safety and Antimicrobial Efficacy of Gel vs. Placebo
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Covid-19 has shut the clinic indefinitely
Sponsor: DermBiont, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: DBI-203
Record Dates: First submitted 2019-12-02; First posted 2019-12-10 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-07

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; S. aureus
MeSH Terms: conditions — Dermatitis, Atopic; Staphylococcal Infections

STUDY DESIGN:
Intervention Model Description: A randomized, observer-blinded, vehicle controlled, single dose application, dose escalating bilateral comparison study of DBI-001 Gel vs. Placebo in the patients with Atopic Dermatitis (AD) affecting the antecubital areas and/or posterior popliteal areas.
  Subjects meeting the inclusion/exclusion criteria and having moderate to heavy growth of S. aureus from a sample collected at screening from an area of dermatitis on at least one arm or at least one leg will be enrolled into the study. Microbiological samples will be collected from all the designated sites on the arms or leg and all subjects will be treated with a single application of the assigned test articles applied by the unblinded treating investigator at the baseline visit.
Who Masked: Outcomes Assessor
Masking Description: This study is Observer Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 DBI-001 Gel and placebo (Active Comparator): Cohort 1 DBI-001 Gel with low dose CFU's of J. lividum and placebo
  Interventions: Drug: J. lividum
- Cohort 2 mid dose DBI-001 Gel and placebo (Active Comparator): Cohort 2 DBI-001 Gel with mid dose CFU's of J. lividum and placebo
  Interventions: Drug: J. lividum
- Cohort 3 high dose DBI-001 Gel and placebo (Active Comparator): Cohort 3 DBI-001 Gel with high dose CFU's of J. lividum. Drug: J. lividum and placebo
  Interventions: Drug: J. lividum

INTERVENTIONS:
Drug: J. lividum — Investigational Product
  Other Names: Janthinobacterium lividum

SUMMARY:
A Randomized, Observer-Blinded, Vehicle Controlled, Single Dose, Dose Escalating, Single Application Within-patient Bilateral Comparison. The goal is to determine the safety and tolerability of DBI-001 Gel vs. Placebo in Adults with Atopic Dermatitis (AD).

DETAILED DESCRIPTION:
A Randomized, Observer-Blinded, Vehicle Controlled, Single Dose, Dose Escalating, Single Application Within-patient Bilateral Comparison. The goal is to determine the safety and tolerability of DBI-001 Gel vs. Placebo in Adults with Atopic Dermatitis and to determine the antibacterial effect of a single application of DBI-001 Gel on the abundance of S. aureus.

Tolerability will be evaluated through assessment of disease state severity and signs and symptoms of local tolerability (pain / burning / stinging, pruritus, erythema, edema, and scabbing / crusting) and review of adverse events. Any local skin reaction that requires use of a concomitant therapy or study discontinuation will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be included in the study:

  1. Ability to understand, agree to, and sign the study Informed Consent. If the patient is unable to provide consent for him/herself, the patient's legally authorized representative may provide written consent.
  2. A signed Health Information Portability and Accountability Act (HIPAA) authorization form which permits the use and disclosure of subject's individually identifiable health information.
  3. Male or Female Subjects of any race 18 years of age and older.
  4. Physician diagnosed clinically stable Atopic Dermatitis according to the criteria of Hanifin and Rajka affecting ≤25% of total BSA with comparable bilateral antecubital or popliteal lesions. Each lesion must have an ADSI ≥6 with a difference between the lesions of ≤1. It will be in the opinion of the Investigator whether the lesions are clinically stable.
  5. Moderate to heavy growth of S. aureus based on culture at the time of screening.
  6. Willingness to discontinue use of other Atopic Dermatitis treatment for the duration of the study unless specifically permitted by the Investigator.
  7. Women of child-bearing potential must:

     * Have negative urine pregnancy tests prior to study treatment to rule out pregnancy, and
     * Use at least one method of birth control that results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner for the duration of study participation.
  8. Willingness not to wash the antecubital lesions on both arms, or the popliteal lesions on both legs, with soap and water from the time of test article application at baseline visit until after the completion of the Day 2 visit.
  9. Allow digital photos of arms or legs to be taken and stored.

Exclusion Criteria:

* 1. Women who are pregnant, planning a pregnancy, or breastfeeding or have a positive pregnancy test at the site.

  2. Any dermatological conditions that could interfere with clinical evaluations or any disease state or physical condition which might expose the patient to an unacceptable risk by study participation.

  3. Any underlying disease(s) or other dermatological conditions that require the use of exclusionary topical or systemic therapy (see Points 5 and 6).

  4. Known sensitivity to any of the components of the study medication. 5. Washout of 4 weeks for topical treatments used on the six designated sites, including but not limited to: antibacterial products, anti-inflammatories (e.g. corticosteroids, tacrolimus, Pimecrolimus). Other than the six sites on the arms or legs, topical mediations may be used before/during the duration of the study.

  6. Willing not to apply any prescription or over the counter topical product on the selected designated sites on arms or legs.

  7. Washout of 4 weeks for systemic treatments for AD, including but not limited to corticosteroids (oral or intramuscular injections), systemic immunomodulators or immunosuppressive (e.g., methotrexate, cyclosporine, hydroxychloroquine), antibiotics (oral or injected, if required to treat a medical condition short duration of oral antibiotics (≤10 days) are permitted after randomization).

  8. Spontaneously improving or rapidly deteriorating dermatitis of the antecubital fossa or popliteal fossa.

  9. Netherton's syndrome or other genodermatoses that result in defective epidermal barrier function.

  10. Washout of 4 weeks for bleach baths. 11. Washout of 4 weeks for phototherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Local Tolerability Based on Scale Listed | Baseline (Day 1) and 14
  Tolerability will be evaluated through assessment of local signs and symptoms. Scoring for burning, stinging, pruritus, erythema, edema, scabbing or crusting. : 0+ none (complete absence), 1=slight (slight), 2=moderate (definitely present), 3=severe (marked, intense).

SECONDARY OUTCOMES:
Change in S. aureus abundance | 14 Days
  Change in the abundance of S. aureus following a single application of DBI-001 Gel.

OTHER OUTCOMES:
Atopic Dermatitis signs and symptoms | 14 Days
  Effect of signs and symptoms of Atopic Dermatitis after a single dose of DBI-001 Gel. • Clinical evaluations will be done by the blinded evaluating investigator of test sites including the Atopic Dermatitis Severity Index (ADSI) and evaluation of erythema, pruritus, exudation, excoriation and lichenification. Scoring: 0+ none (complete absence), 1=slight (slight), 2=moderate (definitely present), 3=severe (marked, intense).

CONTACTS AND LOCATIONS:
Overall Officials: Daisy Blanco, MD, Study Director — Instituto Dermatologico y Cirugia de Piel
Locations (1):
- Instituto Dermatologico y Cirugia de Piel, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No